CLINICAL TRIAL: NCT00730275
Title: A Single-Dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of Sitagliptin in Adolescents
Brief Title: A Study to Assess the Pharmacokinetics, Safety and Tolerability of Sitagliptin in Adolescents (0431-081)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-081; 2008_540
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sitagliptin 50 mg (Experimental): Participants were randomized to sitagliptin 50 mg
  Interventions: Drug: Sitagliptin phosphate
- Sitagliptin 100 mg (Experimental): Participants were randomized to sitagliptin 100 mg
  Interventions: Drug: Sitagliptin phosphate
- Sitagliptin 200 mg (Experimental): Participants were randomized to a single dose of sitagliptin 200 mg
  Interventions: Drug: Sitagliptin phosphate
- Placebo to sitagliptin (Placebo Comparator): Participants were randomized to matching placebo to sitagliptin 50 mg, 100 mg, or 200 mg
  Interventions: Drug: Comparator: matching placebo

INTERVENTIONS:
Drug: Sitagliptin phosphate — Participants will fast 8 hours prior to dosing. All doses will be given with 240 ml of water. Participants received either a single oral dose of sitagliptin 50 mg tablet, sitagliptin 100 mg tablet, or sitagliptin 200 mg.
  Other Names: MK-0431; Januvia
  Arms: Sitagliptin 100 mg; Sitagliptin 200 mg; Sitagliptin 50 mg
Drug: Comparator: matching placebo — Participants will fast 8 hours prior to dosing. All doses will be given with 240 ml of water. Participants received either a single oral dose of matching placebo to sitagliptin 50 mg, 100 mg, or 200 mg.
  Arms: Placebo to sitagliptin

SUMMARY:
This study will assess the safety, tolerability and pharmacokinetics of sitagliptin in 10 to 17 year old diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females who are 10 - 17 years of age
* History of type 2 diabetes
* Nonsmoker
* No clinical or laboratory evidence to indicate a diagnosis of type 1 diabetes

Exclusion Criteria:

* History of diabetic ketoacidosis
* History of stroke, chronic seizures or major neurological disorder
* Consumes alcohol
* Consume more than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola or other beverages containing caffeine per day
* Unable to swallow tablets
* Has had surgery, donated or lost 1 unit of blood, or participated in another investigational study within a minimum of 4 weeks prior to starting the study
* History of multiple and/or severe allergies or has had an allergic reaction to or significant intolerability to prescription or non-prescription drugs or food
* Currently a regular user of any illicit drugs or has a history of drug or alcohol abuse
* History of clinically significant endocrine, gastrointestinal,

cardiovascular, hematological, hepatic, immunological, renal, respiratory, or

genitourinary abnormalities or diseases

* Has an estimated creatinine clearance of less than or equal to 80 mL/min

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2008-07-18 (Actual); Primary Completion 2010-12-30 (Actual); Study Completion 2011-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Fraser IP, Neufeld ND, Fox LA, Kipnes MS, Miller TL, Zeitler PS, Rodriguez H, Gilmartin JH, Lee SJ, Patterson JK, Li XS, Maganti L, Luo WL, Tatosian DA, Stoch SA. A randomized clinical trial to evaluate the single-dose pharmacokinetics, pharmacodynamics, and safety of sitagliptin in pediatric patients with type 2 diabetes. Pediatr Diabetes. 2019 Feb;20(1):48-56. doi: 10.1111/pedi.12790. Epub 2018 Nov 13. PMID 30346099

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin 50 mg: Participants who received a single oral dose of sitagliptin 50 mg.
- Sitagliptin 100 mg: Participants who received a single oral dose of sitagliptin 100 mg.
- Sitagliptin 200 mg: Participants who received a single oral dose of sitagliptin 200 mg.
- Placebo: Participants who received a single oral dose of a matching placebo to sitagliptin 50 mg, 100 mg, or 200 mg.
Period: Overall Study
Arm/Group | Sitagliptin 50 mg | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo
Started | 9 | 9 | 8 | 9
Completed | 9 | 9 | 8 | 8
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 50 mg | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 8 | 9 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.9 (2.52) | 14.3 (1.41) | 14.8 (1.75) | 14.1 (2.26) | 14.3 (1.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 5 | 8 | 24
  Male | 3 | 4 | 3 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Time Frame: Pre-study through 10 to 14 days following administration of study drug
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Sitagliptin 50 mg | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 9
participants | 3 | 1 | 1 | 2

2. Primary Outcome: Area Under the Concentration-time Curve (AUC) From Time 0 to Infinity Following a Single Dose of Sitagliptin
Description: Serum samples were used to determine the AUC from time 0 to infinity for sitagliptin. The placebo group is not included in the table below; this outcome measure only evaluated the sitagliptin groups.
Time Frame: Pre-dose through 72 hours post-dose
Population: All participants who received a single dose of sitagliptin 50 mg, 100 mg, or 200 mg.
Measure: Geometric Mean (95% Confidence Interval); unit: nM*hour
Arm/Group | Sitagliptin 50 mg | Sitagliptin 100 mg | Sitagliptin 200 mg
Number analyzed (Participants) | 9 | 9 | 8
nM*hour | 3438 [2881 to 4103] | 5869 [4918 to 7003] | 12965 [10749 to 15638]

3. Secondary Outcome: Maximum Concentration (Cmax) Following a Single Dose of Sitagliptin
Description: Serum samples were used to determine the Cmax for sitagliptin. The placebo group is not included in the table below; this outcome measure only evaluated the sitagliptin groups.
Time Frame: Pre-dose through 72 hours post-dose
Population: All participants who received a single dose of sitagliptin 50 mg, 100 mg, or 200 mg.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Sitagliptin 50 mg | Sitagliptin 100 mg | Sitagliptin 200 mg
Number analyzed (Participants) | 9 | 9 | 8
nM | 366 [288 to 464] | 666 [526 to 845] | 1876 [1458 to 2413]

4. Secondary Outcome: Time of Occurence of Maximum Concentration (Tmax) Following a Single Dose of Sitagliptin
Description: Serum samples were used to determine the Tmax for sitagliptin. The placebo group is not included in the table below; this outcome measure only evaluated the sitagliptin groups.
Time Frame: Pre-dose through 72 hours post-dose
Population: All participants who received a single dose of sitagliptin 50 mg, 100 mg, or 200 mg.
Measure: Median (Full Range); unit: hours
Arm/Group | Sitagliptin 50 mg | Sitagliptin 100 mg | Sitagliptin 200 mg
Number analyzed (Participants) | 9 | 9 | 8
hours | 3.0 [1.5 to 5.0] | 3.0 [2.0 to 4.5] | 2.5 [1.0 to 3.1]

5. Secondary Outcome: Apparent Terminal Half-life (Apparent t1/2) Following a Single Dose of Sitagliptin
Description: Serum samples were used to determine the apparent t1/2 for sitagliptin. The placebo group is not included in the table below; this outcome measure only evaluated the sitagliptin groups.
Time Frame: Pre-dose through 72 hours post-dose
Population: All participants who received a single dose of sitagliptin 50 mg, 100 mg, or 200 mg.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sitagliptin 50 mg | Sitagliptin 100 mg | Sitagliptin 200 mg
Number analyzed (Participants) | 9 | 9 | 8
hours | 12.1 (1.7) | 11.2 (2.1) | 11.7 (1.8)

6. Secondary Outcome: Plasma Dipeptidyl Peptidase-4 (DPP-4) Activity Following a Single Dose of Sitagliptin or Placebo
Description: Plasma DPP-4 activity was analyzed using the 24-hour weighted average inhibition (WAI) and percent inhibition at 24 hours post-dose.
  WAI was defined as the AUC of inhibition divided by the length of the post-dose time interval. Positive values of WAI represent a decrease in DPP-4 activity.
Time Frame: Pre-dose through 24 hours post-dose
Population: All participants who received a single dose of sitagliptin or placebo.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent inhibition
Groups:
- Placebo: Participants who received a single oral dose of matching placebo to sitagliptin 50 mg, 100 mg, or 200 mg.
Arm/Group | Sitagliptin 50 mg | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 8
Percent inhibition
  24-hour WAI of DPP-4 activity | 73.98 [70.59 to 76.99] | 80.53 [77.98 to 82.78] | 87.96 [86.29 to 89.43] | 6.76 [-6.21 to 18.14]
  DDP-4 activity at 24 hours post-dose | 53.98 [46.74 to 60.24] | 62.78 [56.92 to 67.84] | 75.76 [71.70 to 79.24] | 3.57 [-12.60 to 17.43]

ADVERSE EVENTS:
Arm/Group | Sitagliptin 50 mg | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 3/9 | 1/9 | 1/8 | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 50 mg (N=9) | Sitagliptin 100 mg (N=9) | Sitagliptin 200 mg (N=8) | Placebo (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Infusion site pain (General disorders) | 1 | 0 | 0 | 0
Infusion site swelling (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.